CLINICAL TRIAL: NCT04453722
Title: Wearable Device for Prevention of Opioid-Induced Hypoxemia
Brief Title: Prevention of Opioid-Induced Hypoxemia
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-505; 1R43DA050336-01A1 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-07-01 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Non-cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Monitor only mode: Randomization will be to Oxalert in monitor-only mode
  Interventions: Device: Oxalert Monitor Mode
- Monitor in normal mode: Randomization will be to Oxalert in monitor normal mode which provides progressive audible and tactile alerts for hypoxemia.
  Interventions: Device: Oxalert Normal mode

INTERVENTIONS:
Device: Oxalert Monitor Mode — The investigator will evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO. Using the Oxalert in monitor only mode.
  Groups: Monitor only mode
Device: Oxalert Normal mode — The investigator will evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO using the Oxalert in monitor in normal mode
  Groups: Monitor in normal mode

SUMMARY:
To evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO.

DETAILED DESCRIPTION:
The investigators will evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO. All patients will wear the Oxalert for 24 hours preoperatively in the monitoring only mode (no alerts), throughout hospitalization up to six days, and for 24 post-discharge hours. Randomization will be to Oxalert in monitor-only mode or to its normal mode which provides progressive audible and tactile alerts for hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Adults having major laparoscopic and open abdominal or pelvic surgeries;
* Body Mass Index ≥25 kg/m2
* American Society of Anesthesiologists physical status 1-3;
* Age 18-85 years old;
* Able to understand and consent to the trial and fully participate;
* Anticipated primary opioid analgesia after surgery;
* Expected duration of hospitalization at least 24 hours after surgery;
* Consenting at least 24 hours before anticipated surgery.

Exclusion Criteria:

* Epidural analgesia (field and fascial plane blocks permitted);
* Pre-operative SpO2 <95%;
* No wrist available for the study;
* Severe hearing loss;
* Lack of English language fluency.
* Serious hearing deficit (unable to understand normal speech in a quite environment)
* Serious peripheral neuropathy (unable to feel pin prick at wrist).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll patients who are at increased risk for respiratory insufficiency. Specifically, the investigators will focus on patients scheduled for laparoscopic or open major abdominal or pelvic surgery whose analgesia is primarily opioid-based. The investigators will further restrict enrollment to obese patients (body mass index kg/m2) who are likely to have respiratory compromise. Both men and women will be recruited.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Li K, Saab R, Bravo M, Mascha EJ, Han Y, Nault R, Olson L, Sessler DI. Wearable device for prevention of postoperative and post-discharge hypoxemia: A randomized pilot trial. Acta Anaesthesiol Scand. 2023 Apr;67(4):440-447. doi: 10.1111/aas.14193. Epub 2023 Jan 13. PMID 36583643

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxalert in Monitor Only Mode: Randomization will be to Oxalert in monitor-only mode
  Oxalert Monitor: The investigator will evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO. Using the Oxalert in monitor only mode.
- Oxalert in Monitor in Normal Mode: Randomization will be to Oxalert in monitor normal mode which provides progressive audible and tactile alerts for hypoxemia.
  Oxalert Monitor: The investigator will evaluate the feasibility of a fully randomized validation trial for the Oxalert EPO using the Oxalert in monitor in normal mode
Period: Overall Study
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Started | 24 | 25
Completed | 23 | 24
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12) | 52 (16) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 22 | 21 | 43
  Race: Black | 1 | 4 | 5
  Race: Unknown | 1 | 0 | 1
ASA [Count of Participants; unit: Participants] — Patients were categorized among the 4 ASA physical status according to the pre-anesthesia appointment. This classification uses a grading system of I (better) until IV (worse).
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    mild systemic disease (2) | 6 | 2 | 8
    severe systemic disease (3) | 16 | 21 | 37
    severe systemic disease that is a constant threat to life (4) | 2 | 2 | 4
Surgery type [Count of Participants; unit: Participants]
  Laparoscopy | 6 | 10 | 16
  Open | 18 | 15 | 33
Height [Mean (Standard Deviation); unit: cm] | 170 (10) | 168 (8) | 169 (9)
Weight [Mean (Standard Deviation); unit: kg] | 94 (19) | 92 (16) | 93 (18)
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 32 [28 to 36] | 30 [28 to 38] | 31 [28 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average of SpO2 Below a Threshold of 90%
Description: Time-weighted average of SpO2 below a threshold of 90%. Oxygen Saturation measured between 0% - 100%. Oxygen Saturation <90% is considered abnormal.
Time Frame: during hospitalization up to 6 days and post-discharge 24 hours
Population: number of participants analyzed for in hospital outcome and post-discharge outcome are different
Measure: Median (Inter-Quartile Range); unit: % of SpO2
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 23 | 24
% of SpO2
  In hospital TWA SpO2 <90% (%) | 0.29 [0.04 to 0.71] | 0.11 [0.03 to 0.25]
  Post-discharge TWA SpO2 <90% (%): number analyzed (Participants) | 19 | 19
  Post-discharge TWA SpO2 <90% (%) | 0.16 [0.04 to 0.81] | 0.10 [0.04 to 0.32]
Statistical Analysis 1: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital TWA SpO2 <90% (%); Test type: Superiority — Median difference was estimated from the Hodges-Lehmann estimator of location shift between groups and p-values from Wilcoxon rank sum test; p = 0.120, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0]
Statistical Analysis 2: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital AUC SpO2 <90% (% * min); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.349, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -407, 95% CI 2-sided [-1816 to 208]
Statistical Analysis 3: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Post-discharge TWA SpO2 <90% (%); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.307, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0]
Statistical Analysis 4: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Post-discharge AUC SpO2 <90% (% * min); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.431, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -35, 95% CI 2-sided [-195 to 67]

2. Primary Outcome: Number of Participants With Desaturation Events (Saturation <90%) Lasting at Least 2 Min
Description: Number of Participants with Desaturation Events (Saturation <90%) Lasting at Least 2 Min. All the patients were included.
Time Frame: during hospitalization up to 6 days and post-discharge 24 hours
Population: number of participants analyzed for in hospital outcome and post-discharge outcome are different
Measure: Count of Participants; unit: Participants
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 23 | 24
Participants
  In hospital any event | 20 | 21
  Post-discharge any event: number analyzed (Participants) | 19 | 19
  Post-discharge any event | 14 | 14
Statistical Analysis 1: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital Any event, N (%)c; Test type: Superiority; p > 0.99, Fisher Exact; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.22 to 4.27]
Statistical Analysis 2: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Post-discharge Any event, N (%); Test type: Superiority; p > 0.99, Chi-squared; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.35 to 2.90]

3. Primary Outcome: Duration of Desaturation Events (Saturation <90%) Lasting at Least 2 Min
Description: Duration of Desaturation Events (Saturation <90%) Lasting at Least 2 Mi. All desaturation events were included.
Time Frame: during hospitalization up to 6 days and post-discharge 24 hours
Population: number of participants analyzed for in hospital outcome and post-discharge outcome are different
Measure: Median (Inter-Quartile Range); unit: counts / minutes
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 23 | 24
counts / minutes
  In hospital Total duration | 76 [3 to 531] | 30 [7 to 145]
  In hospital Duration> 2 min | 34 [0.8 to 465] | 8 [2 to 63]
  In hospital Mean duration-all patients | 4.7 [2.8 to 8.6] | 2.7 [2.3 to 3.6]
  In hospital Mean duration for events in those with any events: number analyzed (Participants) | 20 | 21
  In hospital Mean duration for events in those with any events | 5.1 [3.5 to 8.7] | 2.7 [2.6 to 3.7]
  Post-discharge Duration: number analyzed (Participants) | 19 | 19
  Post-discharge Duration | 5 [0 to 70] | 6 [0 to 12]
Statistical Analysis 1: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital Number; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.354, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -6.0, 95% CI 2-sided [-26.0 to 4.0]
Statistical Analysis 2: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital Total duration (min); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.133, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -46.1, 95% CI 2-sided [-274 to 5.1]
Statistical Analysis 3: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital Duration >2 min (min); Test type: Superiority; p = 0.075, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -24.1, 95% CI 2-sided [-213 to 0.1]
Statistical Analysis 4: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: In hospital Mean duration-all patients (min); Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2, 95% CI 2-sided [-4.5 to -0.4]
Statistical Analysis 5: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: in hospital mean duration for events in those with any events (min); Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.2, 95% CI 2-sided [-4.7 to -0.7]
Statistical Analysis 6: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: post-discharge number; Test type: Superiority; p = 0.584, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-4.0 to 1.0]
Statistical Analysis 7: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Post-discharge duration (min); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.556, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.3, 95% CI 2-sided [-18.6 to 3.3]

4. Primary Outcome: AUC of SpO2 Below a Threshold of 90%
Description: AUC of SpO2 Below a Threshold of 90%. SpO2 from 0% -100%.
Time Frame: during hospitalization up to 6 days and post-discharge 24 hours
Measure: Mean (Inter-Quartile Range); unit: % * min
Arm/Group | Monitor Only Mode | Monitor in Normal Mode
Number analyzed (Participants) | 23 | 24
% * min
  In hospital AUC | 1260 [117 to 5278] | 635 [204 to 1513]
  Post-discharge AUC | 130 [47 to 1038] | 121 [27 to 428]

5. Primary Outcome: Number of Desaturation Events (Saturation <90%) Lasting at Least 2 Min
Description: Number of desaturation events (Saturation <90%) Lasting at Least 2 Mi. All desaturation events were included.
Time Frame: during hospitalization up to 6 days and post-discharge 24 hours
Measure: Median (Inter-Quartile Range); unit: counts
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 23 | 24
counts
  In hospital Number | 21 [1 to 69] | 12 [3 to 23]
  Post Discharge Number | 2 [0 to 13] | 2 [0 to 5]

6. Secondary Outcome: Patients' Attitude Toward the Device
Description: We used 0-to-10 (Better - Worst) numerical rating scale to measure the degree of disturbing: 0 = "Not disturbed" and 10 = "Severely disturbed"; others are measured with 5-point numerical rating scales:1="Strongly disagree", 5="Strongly agree" (1=Better - 5= Worst). No subscales combining to compute a total score.
Time Frame: At the day of discharge and after 24 hours of discharge
Population: number of participants analyzed for in hospital outcome and post-discharge outcome are different
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 21 | 21
score on a scale
  Degree of disturbing daily life except sleep (at the day of discharge) | 1.0 [0.0 to 3.0] | 2.0 [1.0 to 4.0]
  Degree of disturbing sleep (at the day of discharge) | 1.0 [0.0 to 1.0] | 2.0 [0.0 to 3.0]
  Comfortable to wear (at the day of discharge) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  Tolerable to audible alert (At the day of discharge): number analyzed (Participants) | 14 | 20
  Tolerable to audible alert (At the day of discharge) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Tolerable to tactile alert (at the day of discharge): number analyzed (Participants) | 8 | 8
  Tolerable to tactile alert (at the day of discharge) | 4.0 [3.0 to 4.0] | 4.0 [3.5 to 4.0]
  Easily cleaned/ disinfected (at the day of discharge): number analyzed (Participants) | 15 | 13
  Easily cleaned/ disinfected (at the day of discharge) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Adequate battery life (at the day of discharge): number analyzed (Participants) | 16 | 19
  Adequate battery life (at the day of discharge) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  Satisfy with the electrode patch (at the day of discharge) | 4.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0]
  Willing to use after study (at the day of discharge) | 4.0 [4.0 to 4.0] | 4.0 [3.0 to 4.0]
  Disturb IV line (at the day of discharge): number analyzed (Participants) | 21 | 19
  Disturb IV line (at the day of discharge) | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Degree of disturbing daily life except sleep (after 24 hours of discharge): number analyzed (Participants) | 20 | 20
  Degree of disturbing daily life except sleep (after 24 hours of discharge) | 2.0 [0.0 to 3.0] | 3.0 [0.50 to 5.0]
  Degree of disturbing sleep (after 24 hours of discharge): number analyzed (Participants) | 20 | 20
  Degree of disturbing sleep (after 24 hours of discharge) | 0.50 [0.00 to 2.5] | 2.0 [0.00 to 4.5]
  Comfortable to wear (after 24 hours of discharge): number analyzed (Participants) | 20 | 20
  Comfortable to wear (after 24 hours of discharge) | 4.0 [3.0 to 4.0] | 3.5 [2.0 to 4.0]
  Tolerable to audible alert (after 24 hours of discharge): number analyzed (Participants) | 13 | 18
  Tolerable to audible alert (after 24 hours of discharge) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Tolerable to tactile alert (after 24 hours of discharge): number analyzed (Participants) | 5 | 9
  Tolerable to tactile alert (after 24 hours of discharge) | 2.0 [2.0 to 4.0] | 4.0 [3.0 to 4.0]
  Easily cleaned/ disinfected (after 24 hours of discharge): number analyzed (Participants) | 18 | 17
  Easily cleaned/ disinfected (after 24 hours of discharge) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Adequate battery life (after 24 hours of discharge): number analyzed (Participants) | 19 | 19
  Adequate battery life (after 24 hours of discharge) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  Satisfy with the electrode patch (after 24 hours of discharge): number analyzed (Participants) | 20 | 20
  Satisfy with the electrode patch (after 24 hours of discharge) | 4.0 [3.5 to 4.0] | 2.5 [2.0 to 4.0]
  Willing to use after study (after 24 hours of discharge): number analyzed (Participants) | 20 | 20
  Willing to use after study (after 24 hours of discharge) | 4.0 [4.0 to 4.0] | 3.5 [3.0 to 4.0]
  Disturb intravenous (IV) line (after 24 hours of discharge): number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Degree of disturbing daily life except sleep (at the day of discharge); Test type: Superiority — Median difference was estimated from the Hodges-Lehmann estimator of location shift between groups and P values from Wilcoxon rank sum test; p = 0.096, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 2.0]
Statistical Analysis 2: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Degree of disturbing sleep (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.205, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 2.0]
Statistical Analysis 3: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: comfortable to wear (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.839, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 4: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Tolerable to audible alert (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.621, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 5: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Tolerable to tactile alert; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.898, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 6: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: easily cleaned/disinfected (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.654, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 7: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: adequate battery life (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.929, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 8: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Satisfy with the electrode patch (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.200, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 9: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Willing to use after study (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.987, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 10: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Disturb IV line (at the day of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.581, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 11: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Degree of disturbing daily life except sleep (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.180, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 3.0]
Statistical Analysis 12: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: degree of distributing sleep (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.171, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 2.0]
Statistical Analysis 13: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Tolerable to audible alert (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.074, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 14: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Tolerable to tactile alert (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.414, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-2.0 to 1.0]
Statistical Analysis 15: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Easily cleaned/disinfected (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.506, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 16: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Adequate battery life (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.747, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 17: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: satisfy with the electrode patch (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.023, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.0]
Statistical Analysis 18: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Willing to use after study (after 24 hours of discharge); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.023, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]

7. Secondary Outcome: Nurses' Attitude Toward the Device
Description: We used 0-to-10 (better- worst) numerical rating scale to measure the degree of disturbing: 0 = "Not disturbed" and 10 = "Severely disturbed"; others are measured with 5-point numerical rating scales:1="Strongly disagree", 5="Strongly agree" (1= better- 5=worst).
Time Frame: Post-operative day 1 (POD 1)
Population: number of participants analyzed for in hospital outcome and post-discharge outcome are different
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
Number analyzed (Participants) | 23 | 25
score on a scale
  Degree of disturbing routine work | 1.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Easily cleaned/ disinfected: number analyzed (Participants) | 13 | 15
  Easily cleaned/ disinfected | 4.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
  Adequate battery life | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 5.0]
  Satisfy with the electrode patch | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 4.0]
  Tolerable to audible alert: number analyzed (Participants) | 4 | 7
  Tolerable to audible alert | 4.0 [3.5 to 4.5] | 4.0 [3.0 to 4.0]
  Willing to use after study | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 5.0]
  Patients' complaint about the device | 2.0 [1.00 to 2.00] | 2.0 [1.0 to 2.0]
  Disturb IV line | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 2.0]
Statistical Analysis 1: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; Degree of disturbing routine work; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.73, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 2: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; Easily cleaned/disinfected; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.097, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 3: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Adequate battery life; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.02, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 4: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Satisfy with the electrode patch; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.037, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 5: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Tolerable to audible alert; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.482, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-2.0 to 1.0]
Statistical Analysis 6: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Willing to use after study; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.031, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 7: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Patients' complaint about the device; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.947, Wilcoxon (Mann-Whitney) — variable: Patients' complaint about the device; Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 8: Comparison: Oxalert in Monitor Only Mode vs Oxalert in Monitor in Normal Mode; variable: Disturb IV line; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.324, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: During hospitalization up to13 days
Arm/Group | Oxalert in Monitor Only Mode | Oxalert in Monitor in Normal Mode
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 3/24 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Oxalert in Monitor Only Mode (N=24) | Oxalert in Monitor in Normal Mode (N=25)
mild blisters on top of Arm after taking off the sticky patch after completing the monitoring part (Skin and subcutaneous tissue disorders) | 1 | 0 — The patient developed mild blisters on top of her Arm after she took off the sticky patch after completing the monitoring part. [MILD]
monitor malfunction (Product Issues) | 1 | 0 — [MILD]
transferred to SICU On POD 1 1/20/2021 due to tachycardia (Cardiac disorders) | 1 | 0 — 010036 transferred to SICU On POD1 1/20/2021 due to tachycardia. IN SICU had a new onset of Atrial fibrillation, , stayed through the last observed day (POD6). [MODERATE]
had 2 episodes of successive tactile and verbal stimulation that caused extreme discomfort (Product Issues) | 0 | 1 — she is convinced that the problem is from the device since she was awake. The first time this happened was in hospital and the second time this happened was at home the night after discharge. [MILD]
Transfer form ward to SICU because of surgical reason (Surgical and medical procedures) | 0 | 1 — [MODERATE]
transferred to SICU On POD 1 1/20/2021 due to shortness of breath and desaturation (Respiratory, thoracic and mediastinal disorders) | 1 | 1/1 — 010036 transferred to SICU On POD1 1/20/2021 due to shortness of breath and desaturation. IN SICU had a new onset of Atrial fibrillation, stayed through the last observed day (POD6).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04453722/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT04453722/ICF_001.pdf